CLINICAL TRIAL: NCT03815838
Title: Molecular Imaging of Pituitary Adenomas
Acronym: MIMOPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cardiff University (Other)
Collaborators: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SPON1592-17
Record Dates: First submitted 2019-01-23; First posted 2019-01-24 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Pituitary Adenoma
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET imaging (Experimental): 18F-FDOPA and 18F-Fallypride PET imaging
  Interventions: Diagnostic Test: PET imaging

INTERVENTIONS:
Diagnostic Test: PET imaging — Positron emission tomography imaging using 18F-Fallypride and 18F-FDOPA
  Other Names: Fallypride; F-DOPA

SUMMARY:
Background: Pituitary adenomas affect 10% of the population. Surgery offers the most cost-effective treatment modality but cure rates are only 40-70%, in part due to the limitations of Magnetic Resonance Imaging (MRI) in visualising small tumours (up to 40% are undetected) and discriminating adenomatous tissue from healthy pituitary or post-surgical change. Positron emission tomography (PET) imaging may improve localisation but current tracers have short half-lives and are unsuitable for routine use. The dopaminergic system regulates pituitary growth and function, as evidenced by the use of dopamine D2 receptor agonists as medical therapy. Dopaminergic PET tracers, including 18F-FDOPA (6-[18F]-L-fluoro-L-3,4-dihydroxyphenylalanine) and 18F (fluorine 18)-Fallypride (which binds to D2/D3 receptors), might thus improve management by enhancing tumour discrimination and quantifying D2 receptor expression.

Aim: To establish whether imaging changes in dopaminergic transmission and receptor function has the potential to improve localisation of pituitary adenomas.

Methods: Subjects with pituitary adenomas will undergo 18F-FDOPA and 18F-Fallypride PET scans in addition to standard pituitary MRI. Quantification of binding potential combined with MRI co-registration to provide enhanced anatomical definition will be applied. In vivo D2 receptor binding will be correlated with ex vivo D2 receptor mRNA (messenger ribonucleic acid) and protein expression from tumour samples removed at surgery.

DETAILED DESCRIPTION:
Aim: In this proof-of-concept study, the investigators will seek to establish whether imaging changes in Dopaminergic transmission and receptor function has the potential to improve localisation and management of pituitary adenomas.

Methods:

Patients will be recruited from the general endocrine and pituitary multidisciplinary clinics at the University Hospital of Wales. Patients will comprise those with a confirmed pituitary adenoma for whom pituitary imaging is indicated as part of standard clinical management. Tumour functionality (Cushing's syndrome, Acromegaly, Prolactinoma, TSHoma) and hypopituitarism will be established in accordance with established clinical practice. Detailed surgical, pathological and post-operative data will be collected in each case, in order to facilitate correlation of PET/MRI findings with key clinical outcomes.

Histopathological examination:

Surgical specimens will be fixed in 10% neutral buffered formalin and embedded in paraffin as per standard clinical practice. Histopathological confirmation of the presence and type of pituitary adenoma will be established by typical microscopic appearances of an adenoma supported by immunohistochemical staining for the relevant hormone (Growth hormone, ACTH [Adrenocorticotrophic Hormone], Prolactin, TSH [Thyroid Stimulating Hormone], LH/FSH [Luteinising hormone/Follicle Stimulating Hormone]). Tumour will also be stored snap frozen for subsequent RNA and protein extraction, in order to quantify dopamine D2 short and long isoform receptor expression. This will allow comparison of ex vivo receptor expression levels with in vivo 18F-fallypride uptake.

PET-CT imaging:

Subjects will undergo 18F-FDOPA and 18F-Fallypride imaging according to established protocols in the PET imaging centre (PETIC) at the University Hospital of Wales. Both compounds will be synthesised in compliance with good manufacturing practice, and have been produced and validated for human use in PETIC since 2015. Subjects will refrain from taking alcohol and caffeine for 4 hours before the PET scanning session. PET scans will be acquired using a PET-CT (Positron Emission Tomography-Computed Tomography) scanner with Time of Flight and a 64 slice CT in 3D list mode. Patients will be placed in the scanner in the supine position, with the brain centred in the axial field of view. A CT scout view will be acquired to aid in positioning of the patient following which the head will be fixed using a piece of surgical tape.

18F-FDOPA protocol: For 18F-FDOPA, participants will be pre-treated with 150 mg (milligrams) carbidopa and 400 mg entacapone 1 hour prior to radioisotope administration in order to block peripheral metabolism of FDOPA and enhance specific signal detection. A low dose CT scan will be acquired for positioning and attenuation correction. A single position Dynamic PET scan will be acquired as 26 time-frames over 94.5 minutes (1 × 30 sec, 4 × 1 min, 3 × 2 min, 3 × 3 min, and 15 × 5 min). Immediately after the scan commences 111 MBq (Megabecquerels) of 18F-DOPA in normal saline will be administered via a long connecting tube as an intravenous bolus at the start of scanning (avoiding brain stimuli). Data will be reconstructed using OSEM (ordered-subsets expectation maximisation) following corrections for attenuation, normalisation, scatter and patient movement. The cerebellum will be used to represent the reference region for the data analysis and enable the generation of binding potential parametric images using Logan plots.

18 F-Fallypride protocol: Dynamic acquisition of the PET scan will be started with a 30 second bolus administration of 18F Fallypride (2.6 MBq/kg body weight). Patients will undergo 3 hours of dynamic imaging (3 × 20 s, 3 × 1 min, 3 × 2 min, 3 × 3 min, 21 × 5 min, 2 × 8 min and 4 × 10 min; 180 min in total)(with rest periods during the scan to reduce discomfort and allow urinary voiding to reduce radiation dose to the bladder wall). Data will be reconstructed using OSEM following corrections for attenuation, normalisation, scatter and patient movement. The cerebellum will be used to represent the reference region for the data analysis and enable the generation of binding potential parametric images using Logan plots.

Standard and 3D gradient echo MRI:

MR imaging will be performed on a 1.5T (Tesla) MRI unit. High resolution coronal T2-weighted images and coronal and sagittal T1-weighted spin echo (SE) images of the pituitary gland will be obtained before contrast injection. After intravenous injection of gadopentetate dimeglumine contrast the investigators will repeat the acquisition of the coronal and sagittal T1-weighted SE images of the pituitary gland and will also record a high resolution T1-weighted spoiled gradient (SPGR) acquisition sequence of the whole head to optimise co-registration with the PET/CT data.

Image processing and analysis:

Image analysis techniques to include detailed profiling of tracer uptake across the sella will be applied. Image processing will be performed using commercially available software packages.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pituitary adenoma for whom pituitary imaging is indicated as part of standard clinical management

Exclusion Criteria:

* Pregnancy, breastfeeding and any contraindications to MRI or intravenous contrast administration

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
PET uptake | 3 hours
  Quantification of tracer binding potential combined with MRI co-registration

CONTACTS AND LOCATIONS:
Overall Officials: Aled Rees, MB BCh, PhD, Principal Investigator — Cardiff University
Locations (1):
- University Hospital of Wales, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No